CLINICAL TRIAL: NCT01776307
Title: A Phase II Clinical Study of BBI608 in Adult Patients With Advanced Colorectal Cancer
Brief Title: A Study of BBI608 in Adult Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBI608-224
Record Dates: First submitted 2013-01-21; First posted 2013-01-28 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
Keywords: BBI608
MeSH Terms: conditions — Colorectal Neoplasms | interventions — napabucasin; Panitumumab; Capecitabine; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BBI608 in combination with cetuximab (Experimental)
  Interventions: Drug: BBI608; Drug: Cetuximab
- BBI608 in combination with panitumumab (Experimental)
  Interventions: Drug: BBI608; Drug: Panitumumab
- BBI608 in combination with capecitabine (Experimental)
  Interventions: Drug: BBI608; Drug: Capecitabine

INTERVENTIONS:
Drug: BBI608 — BBI608 is administered at 500 mg po bid continuously.
  Other Names: Napabucasin; BB608; BBI-608
Drug: Panitumumab — Panitumumab will be administered IV on day 8 and 22 of each 28 day cycle at 6 mg/kg over 60 minutes.
  Other Names: Vectibix
  Arms: BBI608 in combination with panitumumab
Drug: Capecitabine — Capecitabine will be administered orally at 1000 mg/m2 bid daily on days 8-21 every three weeks.
  Other Names: Xeloda
  Arms: BBI608 in combination with capecitabine
Drug: Cetuximab — Cetuximab will be administered IV on day 5 at 400 mg/m2 intravenous infusion over 120 minutes as the initial dose, then weekly at 250mg/m2 over 60-minutes at subsequent cycles.
  Other Names: Erbitux
  Arms: BBI608 in combination with cetuximab

SUMMARY:
This is an open label, multi-center, Phase 2 study of BBI608 in combination with cetuximab, panitumumab or capecitabine in patients with advanced colorectal cancer.

DETAILED DESCRIPTION:
This is an open label, multi-center, Phase 2 study of BBI608 administered in combination with either cetuximab, or panitumumab, or capecitabine. A cycle will consist of daily and continuous oral administration of BBI608 for four weeks in combination with either cetuximab, or panitumumab, or capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent must be obtained and documented according to International Conference on Harmonization (ICH), Good Clinical Practice(GCP), the local regulatory requirements, and permission to use private health information in accordance with the Health Insurance Portability and Accountability Act (HIPPA) prior to study-specific screening procedures.
* A histologically or cytologically confirmed colorectal cancer that is metastatic, unresectable, or recurrent.
* Patients must have received at least 2 regimens containing 5-Fluorouracil,oxaliplatin, or irinotecan.
* Patients to be enrolled in the Cetuximab or Panitumumab combination arms must have colorectal cancer which is K-Ras wild-type.
* ≥ 18 years of age.
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
* Karnofsky performance Status ≥ 70%
* Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last BBI608 dose.
* Females of childbearing potential must have a negative serum pregnancy test.
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤1.5 × upper limit of normal(ULN), or ≤ 2.5 × ULN with metastatic liver disease.
* Hemoglobin (Hgb) ≥ 10 g/dl.
* Total bilirubin ≤ 1.5 × ULN.
* Creatinine ≤ 1.5 × ULN or creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
* Absolute neutrophil count ≥ 1.5 x 10^9/L.
* Platelets ≥ 100 x 10^9/L.
* Life expectancy ≥ 3 months.

Exclusion Criteria:

* Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within four weeks of first dose with the exception for a single dose radiation up to 8 Gray (equal to 800 RAD) with palliative intent for pain control up to 14 days before beginning the administration of BBI608.
* Surgery within 4 weeks prior to first dose.
* Any known symptomatic brain metastases requiring steroids. Patients with treated brain metastases must be stable for 4 weeks after completion of that treatment, with image documentation required. Patients must have no clinical symptoms from brain metastases and must be either off steroids or on a stable dose of steroids for at least 2 weeks prior to protocol enrollment. Patients with known leptomeningeal metastases are excluded, even if treated.
* Pregnant or breastfeeding
* Significant gastrointestinal disorder(s), in the opinion of the Principal Investigator, (e.g., Crohn's disease, ulcerative colitis, extensive gastric and small intestine resection)
* Unable or unwilling to swallow BBI608 capsules daily.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-03; Primary Completion 2018-06 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Edenfield, MD, Principal Investigator — Institute for Translational Oncology Research, Greenville Hospital System
Locations (13):
- United States (13):
  - Mayo Clinic, Scottsdale, Arizona
  - USOR - Rocky Mountain Cancer Center, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - USOR - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - USOR - Northwest Cancer Specialists, Portland, Oregon
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Institute for Translational Oncology Research, Greenville Hospital System, Greenville, South Carolina
  - USOR - Texas Oncology Dallas, Dallas, Texas
  - US Oncology Research, The Woodlands, Texas
  - USOR - Texas Oncology Tyler, Tyler, Texas
  - USOR - Virginia Cancer Specialists, Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 200 participants were enrolled between March 2012 and July 2017.
Pre-assignment Details: Patients who died, withdrew consent to survival follow up or were lost to follow up were considered to have completed the study.
Groups:
- Napabucasin Plus Cetuximab: All participants who were enrolled to Arm A to receive napabucasin administered orally, twice daily in combination with weekly cetuximab administered intravenously
- Napabucasin Plus Panitumumab: All participants who were enrolled to Arm B to receive napabucasin administered orally, twice daily in combination with panitumumab administered intravenously on day 8 and 22 of each 28 day cycle
- Napabucasin Plus Capecitabine: All participants who were enrolled to Arm C to receive napabucasin administered orally, twice daily in combination with capecitabine administered twice daily on days 8-21 every three weeks
Period: Overall Study
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Started | 49 | 75 | 76
Completed | 49 | 75 | 75
Not Completed | 0 | 0 | 1
Not completed — Not dosed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine | Total
Number analyzed (Participants) | 49 | 75 | 75 | 199
Age, Customized [Mean (Standard Deviation); unit: years] | 56.3 (10.37) | 59.7 (11.94) | 58.1 (11.20) | 58.3 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 35 | 24 | 86
  Male | 22 | 40 | 51 | 113
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 8 | 14
  White | 39 | 69 | 64 | 172
  More than one race | 3 | 2 | 0 | 5
  Unknown or Not Reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate
Description: Assessment of Disease Control Rate, defined as the proportion of patients with a documented complete response, partial response and stable disease based on RECIST 1.1, in patients with advanced colorectal cancer given napabucasin in combination with cetuximab, panitumumab or capecitabine
Time Frame: From the date of first treatment, every 8 weeks, until the date of first documented objective disease progression, up to 24 months
Population: Patients who received at least 1 cycle of study treatment and had at least 1 disease assessment following the initiation of therapy. Patients missing imaging assessment following the initiation of treatment are not included in the assessment for DCR.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Napabucasin Plus Cetuximab: Napabucasin administered orally, twice daily, in combination with weekly cetuximab administered intravenously on Days 5, 12, 19, and 26 of each 28 day study cycle. Patients in this group had a baseline scan and at least one assessment approximately 8 weeks from baseline.
- Napabucasin Plus Panitumumab: Napabucasin administered orally, twice daily, in combination with panitumumab administered intravenously on Days 8 and 22 of each 28 day study cycle. Patients in this group had a baseline scan and at least one assessment approximately 8 weeks from baseline.
- Napabucasin Plus Capecitabine: Napabucasin administered orally, twice daily, in combination with capecitabine administered twice daily on Days 8-21 every three weeks. Patients in this group had a baseline scan and at least one assessment approximately 8 weeks from baseline.
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 29 | 41 | 39
Percentage of participants | 34.5 [17.9 to 54.3] | 36.6 [22.1 to 53.1] | 25.6 [13.0 to 42.1]
Statistical Analysis 1: Comparison: Napabucasin Plus Cetuximab vs Napabucasin Plus Panitumumab vs Napabucasin Plus Capecitabine; Test type: Other — Descriptive analysis for investigational arms; no comparator analysis; The exact 95% confidence interval is based on the Clopper-Pearson method

2. Secondary Outcome: Progression Free Survival
Description: The effect of napabucasin given in combination with cetuximab, panitumumab or capecitabine on Progression Free Survival (PFS) of patients with advanced colorectal cancer.
Time Frame: The time from the date of first treatment to the date of first documentation of disease progression or death due to any cause, up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Napabucasin Plus Cetuximab: Napabucasin administered orally, twice daily, in combination with weekly cetuximab administered intravenously on Days 5, 12, 19, and 26 of each 28 day study cycle . Patients in this group had a baseline scan and at least one on study scan or died from any cause.
- Napabucasin Plus Panitumumab: Napabucasin administered orally, twice daily, in combination with panitumumab administered intravenously on Days 8 and 22 of each 28 day study cycle. Patients in this group had a baseline scan and at least one on study scan or died from any cause.
- Napabucasin Plus Capecitabine: Napabucasin administered orally, twice daily, in combination with capecitabine administered twice daily on Days 8-21 every three weeks. Patients in this group had a baseline scan and at least one on study scan or died from any cause
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 49 | 75 | 75
months | 1.87 [1.81 to 3.65] | 2.27 [2.04 to 3.58] | 1.94 [1.71 to 2.73]
Statistical Analysis 1: Comparison: Napabucasin Plus Cetuximab vs Napabucasin Plus Panitumumab vs Napabucasin Plus Capecitabine; Test type: Other — Estimates provided for investigational arms; no comparator analysis; Estimated from Kaplan Meier Curve

3. Secondary Outcome: Overall Survival
Description: The effect of napabucasin given in combination with cetuximab, panitumumab or capecitabine on the Overall Survival of patients with advanced colorectal cancer
Time Frame: 4 weeks after the patient has been off study treatment, every 3 months thereafter until death, up to 60 months.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Napabucasin Plus Cetuximab: Napabucasin administered orally, twice daily, in combination with weekly cetuximab administered intravenously on Days 5, 12, 19, and 26 of each 28 day study cycle.
- Napabucasin Plus Panitumumab: Napabucasin administered orally, twice daily, in combination with panitumumab administered intravenously on Days 8 and 22 of each 28 day study cycle.
- Napabucasin Plus Capecitabine: Napabucasin administered orally, twice daily, in combination with capecitabine administered twice daily on Days 8-21 every three weeks.
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 49 | 75 | 75
Months | 7.79 [5.49 to 8.54] | 9.10 [5.88 to 12.48] | 6.34 [5.13 to 11.33]
Statistical Analysis 1: Comparison: Napabucasin Plus Cetuximab vs Napabucasin Plus Panitumumab vs Napabucasin Plus Capecitabine; Test type: Other — Estimates provided for investigational arms; no comparator analysis; Estimated from Kaplan Meier Curve

4. Secondary Outcome: Determination of the Maximum Observed Concentration (Cmax) of Napabucasin When Administered 480mg, Twice Daily, on Day 5 of the First Study Cycle
Description: To determine the maximum concentration of napabucasin when given at 480mg, twice daily, in combination with cetuximab, panitumumab, or capecitabine in patients with advanced colorectal cancer.
Time Frame: Blood samples drawn on day 5 during the first study cycle
Population: Napabucasin plus capecitabine: No evaluable patients dosed at 480mg twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Napabucasin Plus Cetuximab: Napabucasin administered orally, twice daily, in combination with weekly cetuximab administered intravenously on Days 5, 12, 19, and 26 of each 28 day study cycle. Patients included in this group took napabucasin 480mg twice daily and provided blood samples for analysis.
- Napabucasin Plus Panitumumab: Napabucasin administered orally, twice daily, in combination with panitumumab administered intravenously on Days 8 and 22 of each 28 day study cycle. Patients included in this group took napabucasin 480mg twice daily and provided blood samples for analysis.
- Napabucasin Plus Capecitabine: Napabucasin administered orally, twice daily, in combination with capecitabine administered twice daily on Days 8-21 every three weeks. Patients included in this group took napabucasin 480mg twice daily and provided blood samples for analysis.
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 6 | 1 | 0
ng/mL | 661 (77.9) | 468 (NA) — Not calculated |

5. Secondary Outcome: Determination of the Maximum Observed Concentration (Cmax) of Napabucasin When Administered 480mg, Twice Daily, on Day 21 of the First Study Cycle
Description: as for outcome 4
Time Frame: Blood samples drawn on day 21 during the first study cycle
Population: Napabucasin plus capecitabine: No evaluable patients dosed at 480mg twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 5 | 1 | 0
ng/mL | 627 (77.3) | 398 (NA) — Not calculated |

6. Secondary Outcome: Determination of the Maximum Observed Concentration (Cmax) of Napabucasin When Administered 240mg, Twice Daily, on Day 21 of the First Study Cycle
Description: To determine the maximum concentration of napabucasin when given at 240mg, twice daily, in combination with cetuximab, panitumumab, or capecitabine in patients with advanced colorectal cancer.
Time Frame: Blood samples drawn on day 21 during the first study cycle
Population: Napabucasin plus panitumumab & Napabucasin plus capecitabine: No evaluable patients dosed at 240mg twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Napabucasin Plus Cetuximab: Napabucasin administered orally, twice daily, in combination with weekly cetuximab administered intravenously on Days 5, 12, 19, and 26 of each 28 day study cycle. Patients included in this group took napabucasin 240mg twice daily and provided blood samples for analysis.
- Napabucasin Plus Panitumumab: Napabucasin administered orally, twice daily, in combination with panitumumab administered intravenously on Days 8 and 22 of each 28 day study cycle. Patients included in this group took napabucasin 240mg twice daily and provided blood samples for analysis.
- Napabucasin Plus Capecitabine: Napabucasin administered orally, twice daily, in combination with capecitabine administered twice daily on Days 8-21 every three weeks. Patients included in this group took napabucasin 240mg twice daily and provided blood samples for analysis.
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 1 | 0 | 0
ng/mL | 494 (NA) — Not calculated |  |

7. Secondary Outcome: Determination of the Maximum Observed Concentration (Cmax) of Napabucasin When Administered 500mg, Twice Daily, on Day 5 of the First Study Cycle
Description: To determine the maximum concentration of napabucasin when given at 500mg, twice daily, in combination with cetuximab, panitumumab, or capecitabine in patients with advanced colorectal cancer.
Time Frame: Blood samples drawn on day 5 during the first study cycle
Population: Napabucasin plus cetuximab: No evaluable patients dosed at 500mg twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Napabucasin Plus Cetuximab: Napabucasin administered orally, twice daily, in combination with weekly cetuximab administered intravenously on Days 5, 12, 19, and 26 of each 28 day study cycle. Patients included in this group took napabucasin 500mg twice daily and provided blood samples for analysis.
- Napabucasin Plus Panitumumab: Napabucasin administered orally, twice daily, in combination with panitumumab administered intravenously on Days 8 and 22 of each 28 day study cycle. Patients included in this group took napabucasin 500mg twice daily and provided blood samples for analysis.
- Napabucasin Plus Capecitabine: Napabucasin administered orally, twice daily, in combination with capecitabine administered twice daily on Days 8-21 every three weeks. Patients included in this group took napabucasin 500mg twice daily and provided blood samples for analysis.
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 0 | 4 | 6
ng/mL |  | 1020 (50.6) | 858 (34.5)

8. Secondary Outcome: Determination of the Maximum Observed Concentration (Cmax) of Napabucasin When Administered 500mg, Twice Daily, on Day 21 of the First Study Cycle
Description: as for outcome 7
Time Frame: Blood samples drawn on day 21 during the first study cycle
Population: Napabucasin plus cetuximab: No evaluable patients dosed at 500mg twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 0 | 3 | 5
ng/mL |  | 1060 (23.0) | 789 (72.0)

9. Secondary Outcome: Area Under the Plasma Concentration vs. Time Curve (AUClast) of Napabucasin When Administered 480mg, Twice Daily, on Day 5 of the First Study Cycle
Description: To determine the area under the plasma concentration vs. time curve of napabucasin when given at 480mg, twice daily, in combination with cetuximab, panitumumab, or capecitabine in patients with advanced colorectal cancer.
Time Frame: Blood samples drawn on day 5 during the first study cycle
Population: Napabucasin plus capecitabine: No evaluable patients dosed at 480mg twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 6 | 1 | 0
h*ng/mL | 3380 (83.3) | 2730 (NA) — Not calculated |

10. Secondary Outcome: Area Under the Plasma Concentration vs. Time Curve (AUClast) of Napabucasin When Administered 480mg, Twice Daily, on Day 21 of the First Study Cycle
Description: as for outcome 9
Time Frame: Blood samples drawn on day 21 during the first study cycle
Population: Napabucasin plus capecitabine: No evaluable patients dosed at 480mg twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 5 | 1 | 0
h*ng/mL | 2930 (137) | 2630 (NA) — Not calculated |

11. Secondary Outcome: Area Under the Plasma Concentration vs. Time Curve (AUClast) of Napabucasin When Administered 240mg, Twice Daily, on Day 21 of the First Study Cycle
Description: To determine the area under the plasma concentration vs. time curve of napabucasin when given at 240mg, twice daily, in combination with cetuximab, panitumumab, or capecitabine in patients with advanced colorectal cancer.
Time Frame: Blood samples drawn on day 21 during the first study cycle
Population: Napabucasin plus panitumumab and Napabucasin plus capecitabine: No evaluable patients dosed at 240mg twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 1 | 0 | 0
h*ng/mL | 2870 (NA) — Not calculated |  |

12. Secondary Outcome: Area Under the Plasma Concentration vs. Time Curve (AUClast) of Napabucasin When Administered 500mg, Twice Daily, on Day 5 of the First Study Cycle
Description: To determine the area under the plasma concentration vs. time curve of napabucasin when given at 500mg, twice daily, in combination with cetuximab, panitumumab, or capecitabine in patients with advanced colorectal cancer.
Time Frame: Blood samples drawn on day 5 during the first study cycle
Population: Napabucasin plus cetuximab: No evaluable patients dosed at 500mg twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 0 | 4 | 6
h*ng/mL |  | 5420 (36.3) | 5350 (38.7)

13. Secondary Outcome: Area Under the Plasma Concentration vs. Time Curve (AUClast) of Napabucasin When Administered 500mg, Twice Daily, on Day 21 of the First Study Cycle
Description: as for outcome 12
Time Frame: Blood samples drawn on day 21 during the first study cycle
Population: Napabucasin plus cetuximab: No evaluable patients dosed at 500mg twice daily.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 0 | 3 | 5
h*ng/mL |  | 6290 (6.71) | 4720 (48.2)

14. Secondary Outcome: Pharmacodynamics
Description: To determine the response (increase or decrease) of biomarkers from biopsied tumors following the administration of napabucasin
Time Frame: During the first 28 days of the study cycle
Population: No on-treatment biopsies were performed therefore no pharmacodynamic testing on tumor tissue was conducted.
Groups:
- Napabucasin Plus Cetuximab: Napabucasin administered orally, twice daily, in combination with weekly cetuximab administered intravenously on Days 5, 12, 19, and 26 of each 28 day study cycle . Patients included in this group needed to have on treatment biopsy
- Napabucasin Plus Panitumumab: Napabucasin administered orally, twice daily, in combination with panitumumab administered intravenously on Days 8 and 22 of each 28 day study cycle. Patients included in this group needed to have on treatment biopsy
- Napabucasin Plus Capecitabine: Napabucasin administered orally, twice daily, in combination with capecitabine administered twice daily on Days 8-21 every three weeks. Patients included in this group needed to have on treatment biopsy.
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Number of Patients With Adverse Events and Serious Adverse Events
Description: Assessment of safety of napabucasin given in combination with cetuximab, panitumumab or capecitabine to patients with advanced colorectal cancer by reporting of adverse events and serious adverse events
Time Frame: The time from the date of first treatment, while the patient is taking napabucasin, and for 30 days after stopping therapy, an average of 4 months.
Measure: Count of Participants; unit: Participants
Groups:
- Napabucasin Plus Cetuximab: Napabucasin administered orally, twice daily, in combination with weekly cetuximab administered intravenously on Days 5, 12, 19, and 26 of each 28 day study cycle. Patients included in this group received at least one dose of study drug.
- Napabucasin Plus Panitumumab: Napabucasin administered orally, twice daily, in combination with panitumumab administered intravenously on Days 8 and 22 of each 28 day study cycle. Patients included in this group received at least one dose of study drug.
- Napabucasin Plus Capecitabine: Napabucasin administered orally, twice daily, in combination with capecitabine administered twice daily on Days 8-21 every three weeks. Patients included in this group received at least one dose of study drug.
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
Number analyzed (Participants) | 49 | 75 | 75
Participants | 49 | 75 | 75

ADVERSE EVENTS:
Time Frame: Serious and Other Adverse Events were assessed from the date of first treatment through 30 days of the last administration of study drug, an average of 4 months. All-Cause Mortality was assessed from the date of first treatment until death, assessed up to 60 months.
Groups:
- Napabucasin Plus Cetuximab: All participants who received at least 1 dose of napabucasin administered orally, twice daily in combination with weekly cetuximab administered intravenously
- Napabucasin Plus Panitumumab: All participants who received at least 1 dose of napabucasin administered orally, twice daily in combination with panitumumab administered intravenously on day 8 and 22 of each 28 day cycle
- Napabucasin Plus Capecitabine: All participants who received at least 1 dose of napabucasin administered orally, twice daily in combination with capecitabine administered twice daily on days 8-21 every three weeks
Arm/Group | Napabucasin Plus Cetuximab | Napabucasin Plus Panitumumab | Napabucasin Plus Capecitabine
All-Cause Mortality (participants affected / at risk) | 45/49 | 70/75 | 72/75
Serious Adverse Events (participants affected / at risk) | 17/49 | 29/75 | 26/75
Other Adverse Events (participants affected / at risk) | 49/49 | 75/75 | 75/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Napabucasin Plus Cetuximab (N=49) | Napabucasin Plus Panitumumab (N=75) | Napabucasin Plus Capecitabine (N=75)
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 4 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2
Ascites (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Disease progression (General disorders) | 3 | 3 | 0
Pyrexia (General disorders) | 0 | 3 | 0
Chest pain (General disorders) | 0 | 1 | 0
Device dislocation (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 3
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 3
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Renal haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Napabucasin Plus Cetuximab (N=49) | Napabucasin Plus Panitumumab (N=75) | Napabucasin Plus Capecitabine (N=75)
Diarrhoea (Gastrointestinal disorders) | 37 | 58 | 61
Abdominal pain (Gastrointestinal disorders) | 25 | 26 | 30
Nausea (Gastrointestinal disorders) | 22 | 39 | 47
Vomiting (Gastrointestinal disorders) | 22 | 27 | 27
Constipation (Gastrointestinal disorders) | 15 | 9 | 10
Abdominal pain upper (Gastrointestinal disorders) | 6 | 6 | 7
Ascites (Gastrointestinal disorders) | 2 | 5 | 3
Abdominal distension (Gastrointestinal disorders) | 3 | 3 | 6
Stomatitis (Gastrointestinal disorders) | 1 | 5 | 4
Decreased appetite (Metabolism and nutrition disorders) | 15 | 24 | 23
Hypomagnesaemia (Metabolism and nutrition disorders) | 15 | 23 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 23 | 15
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 8 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 7 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 2 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 15 | 22
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 5 | 2
Hypouricaemia (Metabolism and nutrition disorders) | 10 | 4 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 10 | 13 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 9 | 21 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 9 | 1
Palmar-plantar erythrodysaethesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 5 | 11
Fatigue (General disorders) | 20 | 43 | 36
Oedema peripheral (General disorders) | 6 | 6 | 8
Pyrexia (General disorders) | 6 | 5 | 7
Mucosal inflammation (General disorders) | 5 | 3 | 3
Chills (General disorders) | 3 | 6 | 3
Disease progression (General disorders) | 3 | 3 | 0
Asthenia (General disorders) | 0 | 5 | 7
Dizziness (Nervous system disorders) | 7 | 7 | 9
Headache (Nervous system disorders) | 5 | 6 | 3
Chromaturia (Renal and urinary disorders) | 11 | 12 | 10
Proteinuria (Renal and urinary disorders) | 5 | 11 | 18
Ketonuria (Renal and urinary disorders) | 3 | 11 | 17
Haematuria (Renal and urinary disorders) | 2 | 9 | 10
Glycosuria (Renal and urinary disorders) | 0 | 2 | 6
Anaemia (Blood and lymphatic system disorders) | 9 | 16 | 16
Lymphopenia (Blood and lymphatic system disorders) | 1 | 9 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 6 | 5
Leukopenia (Blood and lymphatic system disorders) | 1 | 4 | 5
Blood alkaline phosphatase increased (Investigations) | 7 | 9 | 12
Aspartate aminotransferase increased (Investigations) | 6 | 6 | 13
Blood bilirubin increased (Investigations) | 4 | 6 | 1
Alanine aminotransferase increased (Investigations) | 4 | 5 | 5
Blood lactate dehydrogenase increased (Investigations) | 4 | 1 | 0
Blood creatinine increased (Investigations) | 3 | 1 | 5
Weight decreased (Investigations) | 1 | 5 | 5
Protein total decreased (Investigations) | 0 | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 13 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 9 | 10
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5
Urinary tract infection (Infections and infestations) | 4 | 15 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 4 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4
Vision blurred (Eye disorders) | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 3 | 3
Anxiety (Psychiatric disorders) | 3 | 3 | 3
Depression (Psychiatric disorders) | 1 | 5 | 4
Hypotension (Vascular disorders) | 3 | 4 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and embargo communications of results up to 60 days.

DOCUMENTS (2):
  • Study Protocol (2014-10-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT01776307/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT01776307/SAP_001.pdf